CLINICAL TRIAL: NCT05653427
Title: A Phase 2, Open-Label Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Amivantamab Monotherapy in Participants With Previously Treated Advanced Hepatocellular Carcinoma
Brief Title: A Study of Amivantamab Monotherapy in Participants With Previously Treated Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: N~15 subjects data analysis did not meet statistical consideration of ORR and study primary/secondary objectives were not met. Enrollment was terminated for futility
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109249; 61186372HCC2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Amivantamab Monotherapy (Experimental): Participants will receive amivantamab monotherapy intravenously once weekly on Days 1 and 2 in Cycle 1 and on Days 1 and 15 from Cycle 2 onwards based on body weight. Each cycle is of 28 days.
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered intravenously.
  Other Names: JNJ-61186372

SUMMARY:
The purpose of this study is to characterize the preliminary antitumor activity of amivantamab at the recommended dose in participants with previously systemically treated hepatocellular carcinoma (HCC)

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed diagnosis of hepatocellular carcinoma (HCC) (fibrolamellar and mixed hepatocellular / cholangiocarcinoma subtypes are not eligible) based on pathology report, who have barcelona clinic liver cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach
* Participant must have measurable disease according to response criteria in solid tumors (RECIST) Version 1.1. Selected target lesions must meet 1 of 2 criteria: 1) not previously treated with local therapy or 2) within the field of prior local therapy but with documented subsequent progression as per RECIST v1.1
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Participant must have adequate organ and bone marrow function
* A female participant must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 6 months after receiving the last dose of study treatment. Female participants should consider preservation of eggs prior to study treatment as anti-cancer treatments may impair fertility

Exclusion Criteria:

* Participants with prior liver transplant, history of hepatic encephalopathy, portal vein invasion at the main portal branch (Vp4), inferior vena cava, or cardiac involvement of HCC based on imaging, or any current moderate or severe ascites as measured by physical examination that requires active paracentesis for control due to the underlying HCC
* Participant has known allergies, hypersensitivity, or intolerance to excipients of amivantamab
* Participant has received a live or live attenuated vaccine within 3 months before Cycle 1 Day 1. The seasonal influenza vaccine and non-live vaccines against Coronavirus disease 19 (COVID-19) are not exclusionary
* Other clinically active liver disease of infectious origin
* Participant has a history of clinically significant cardiovascular disease including, but not limited to: a. diagnosis of deep vein thrombosis or pulmonary embolism within 4 weeks prior to the first dose of study treatment or any of the following within 6 months prior to the first dose of study treatment: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome. Clinically non-significant thrombosis, such as nonobstructive catheter-associated clots, are not exclusionary; b. prolonged corrected QT interval using Fridericia's formula (QTcF) greater than (>)480 millisecond (msec) or clinically significant cardiac arrhythmia or electrophysiologic disease (example, placement of implantable cardioverter defibrillator or atrial fibrillation with uncontrolled rate); c. uncontrolled (persistent) hypertension: systolic blood pressure >160 mm Hg; diastolic blood pressure >100 millimeter of mercury (mm Hg), or congestive heart failure (CHF) defined as New York Heart Association (NYHA) class III/IV or hospitalization for CHF (any NYHA class) within 6 months of study enrollment; d. pericarditis/clinically significant pericardial effusion; e. myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- China (13):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Chang Chun Shi
  - The Third Xiangya Hospital, Central South University, Changsha
  - West China Hospital, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou
  - Nanfang Hospital, Guangzhou
  - Zhejiang University First Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Second Affiliatde Hospital To Nanchang University, Nanchang
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Xi An International Medical Center Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 3 parts: Part 1, main Part 2 and expansion Part 3. However, due to the early termination of study, the enrollment was discontinued before planned enrollment was achieved in Part 2. Due to changes in the planned analysis, efficacy and safety data were analyzed together for Part 1 and Part 2 and Part 3 was not conducted. As a result, combined results for both parts were presented.
Groups:
- Amivantamab Monotherapy (1050/1400 mg): Participants with previously treated advanced hepatocellular carcinoma (HCC) received amivantamab 1050 milligrams (mg) for body weight less than (<) 80 kilograms (kg) or 1400 mg for body weight greater than or equal to (>=) 80 kg as an intravenous (IV) infusion in each 28-day cycles. During Cycle 1, amivantamab was administered once weekly on Days 1, 8, 15 and 22 with first dose split over Day 1 (350 mg) and Day 2 (700 mg for body weight <80 kg/1050 mg for body weight >=80 kg). From Cycle 2 onwards, amivantamab was administered on Days 1 and 15 until documented clinical or radiographic disease progression or until the participant discontinued study treatment due to withdrawal of consent, safety reasons, noncompliance with study drug administration or procedural requirements with treatment continuing for a maximum of up to 2.8 months. Participants were followed up for safety every 12 weeks after the last dose of study treatment or disease progression until the end of study, death, lost to follow-up, or withdrawal of consent, whichever comes first.
Period: Overall Study
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Started | 18
Completed | 5
Not Completed | 13
Not completed — Study Terminated by Sponsor | 13

BASELINE CHARACTERISTICS:
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  CHINA | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 by Investigator Assessment
Description: ORR was defined as the percentage of participants who achieved a confirmed complete response (CR) or partial response (PR) as determined by investigator per RECIST version 1.1. As per RECIST version 1.1, CR was defined as disappearance of all extranodal lesions, the regression of all nodal lesions to less than (<)10 millimeter (mm) short axis and the normalization of tumor marker level. PR was defined as greater than or equal to (>=) 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference baseline sum of diameters of target lesions.
Time Frame: From start of treatment on Day 1 up to 3.8 months
Population: Response evaluable analysis set included all participants who received at least 1 dose of study treatment; had at least 1 post-baseline efficacy disease assessment, or discontinued treatment for any reason, or had disease progression/death prior to the first post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Percentage of participants | 0.0 [0.0 to 18.5]

2. Secondary Outcome: Duration of Response (DOR) as Per RECIST Version 1.1
Description: DOR was defined as time from date of first documented response (CR/PR) until date of first documented progressive disease (PD) or death, whichever occurred first. As per RECIST version 1.1, CR was defined as disappearance of all extranodal lesions, the regression of all nodal lesions to <10 mm short axis and the normalization of tumor marker level. PR was defined as >=30% decrease in the sum of diameters of target lesions, taking as reference baseline sum of diameters of target lesions. PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started. There was no participant who had event (CR/PR), hence data could not be collected and analyzed for this outcome measure.
Time Frame: From the date of first documented response up to date of first documented PD or death (up to 3.8 months)
Population: Response evaluable analysis set included all participants who received at least 1 dose of study treatment; had at least 1 post-baseline efficacy disease assessment, or discontinued treatment for any reason, or had disease progression/death prior to the first post-baseline disease assessment. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease Control Rate (DCR) as Per RECIST Version 1.1
Description: DCR was defined as the percentage of participants achieving CR or PR or stable disease (SD) for at least 11 weeks as defined by RECIST version 1.1. As per RECIST version 1.1, CR was defined as disappearance of all extranodal lesions, the regression of all nodal lesions to <10 mm short axis and the normalization of tumor marker level. PR was defined as >=30% decrease in the sum of diameters of target lesions, taking as reference baseline sum of diameters of target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started.
Time Frame: From start of treatment on Day 1 up to 3.8 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Percentage of participants | 0.0 [0.0 to 18.5]

4. Secondary Outcome: Progression Free Survival (PFS) as Per RECIST Version 1.1
Description: PFS was defined as the time from the date of first dose of study drug until the date of objective disease progression or death by any cause, whichever comes first, based on investigator assessment using RECIST Version 1.1. PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started.
Time Frame: From start of the treatment (Day 1) until disease progression or death (up to 3.8 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Months | 1.48 [1.41 to 1.51]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study drug until the date of death due to any cause.
Time Frame: From start of the treatment (Day 1) until death due to any cause (up to 3.8 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Months | NA [3.84 to NA] — Here, 'NA' signifies that median and upper limit of 95% confidence interval (CI) could not be calculated due to less number of participants with events.

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs was defined as AEs occurring at or after first dose of study drug up to 30 days after last dose or until the start of new anticancer therapy, whichever occurred first. TEAEs were graded according to NCI-CTCAE version 5.0. Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe or medically significant but not immediately life-threatening; Grade 4- Life-threatening consequences; Grade 5- Death related to AE. All TEAEs including serious and non-serious events were reported in this outcome measure.
Time Frame: From start of the treatment (Day 1) up to 30 days after last dose of study drug or start of subsequent anticancer therapy (up to 3.8 months)
Population: All treated analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Participants
  Grade 1 | 5
  Grade 2 | 9
  Grade 3 | 3
  Grade 4 | 0
  Grade 5 | 1

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Number of participants with clinically significant abnormalities in laboratory parameters (serum chemistry and hematology) were reported. Clinically significant abnormalities were determined based on investigator's discretion.
Time Frame: as for outcome 6
Population: All treated analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Participants | 3

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs Values
Description: Vital signs assessments included systolic and diastolic blood pressure, heart rate, respiratory rate, pulse rate, body temperature and oxygen saturation. These measurements were taken after the participants had rested for at least 5 minutes in a quiet setting without distractions. Clinical significance of any vital signs was determined based on investigator's discretion.
Time Frame: as for outcome 6
Population: All treated analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 18
Participants | 0

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Amivantamab
Description: Cmax was defined as the maximum observed serum concentration of amivantamab. The concentrations of amivantamab were measured using a validated, specific, and sensitive enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Pre-dose, 0, 24, 26, 30, 48, 96 and 168 hours post-dose on Day 1 of Cycle 1; pre-dose, 0, 2, 6, 24, 72, 168, 240 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: Pharmacokinetics (PK) analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable postbaseline measurement. Here 'N' (overall number of participants analyzed) refers to the participants evaluable for this outcome measure and 'n' (number analyzed) refers to the participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (mcg/mL)
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 5
Micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1 | 339 (57.0)
  Cycle 2 Day 1: number analyzed (Participants) | 4
  Cycle 2 Day 1 | 711 (79.0)

10. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of Amivantamab
Description: Tmax was defined as the time to reach maximum observed serum concentration of amivantamab. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: as for outcome 9
Population: PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable postbaseline measurement. Here 'N' (overall number of participants analyzed) refers to the participants evaluable for this outcome measure and 'n' (number analyzed) refers to the participants evaluable at specified time points.
Measure: Median (Full Range); unit: Hours
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 5
Hours
  Cycle 1 Day 1 | 27.18 [25.68 to 28.70]
  Cycle 2 Day 1: number analyzed (Participants) | 4
  Cycle 2 Day 1 | 5.87 [2.27 to 7.75]

11. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Time 168 Hours (h) (AUC [0-168h]) of Amivantamab
Description: AUC (0-168h) was defined as area under the serum concentration time-curve from time zero to the time point 168 hours. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: Pre-dose, 0, 24, 26, 30, 48, 96 and 168 hours post-dose on Day 1 of Cycle 1; pre-dose, 0, 2, 6, 24, 72 and 168 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: micrograms*hours/milliliter (mcg*hr/mL)
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 5
micrograms*hours/milliliter (mcg*hr/mL)
  Cycle 1 Day 1 | 29084 (3772)
  Cycle 2 Day 1: number analyzed (Participants) | 4
  Cycle 2 Day 1 | 80434 (11319)

12. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to End of Dosing Interval (AUCtau) of Amivantamab
Description: Area under the serum concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval of 336 hours was reported. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: Pre-dose, 0, 2, 6, 24, 72, 168, 240 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable postbaseline measurement. Here 'N' (overall number of participants analyzed) refers to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 3
mcg*hr/mL | 117913 (19426)

13. Secondary Outcome: Serum Trough Concentrations (Ctrough) of Amivantamab: on Days 8 and 15 of Cycle 1; Day 1 of Cycle 2 and Cycle 4; Day 15 of Cycle 2 and Cycle 3
Description: Ctrough of amivantamab at pre-dose on Days 8 and 15 of Cycle 1; Day 1 of Cycle 2 and Cycle 4; Day 15 of Cycle 2 and Cycle 3 were reported. Ctrough was defined as pre-dose serum drug concentration. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: Pre-dose at 0 hour: Days 8 and 15 of Cycle 1; Day 1 of Cycle 2 and Cycle 4; Day 15 of Cycle 2 and Cycle 3 (each cycle was of 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 17
mcg/mL
  Pre-dose Cycle 1 Day 8 | 145 (103)
  Pre-dose Cycle 1 Day 15: number analyzed (Participants) | 16
  Pre-dose Cycle 1 Day 15 | 229 (117)
  Pre-dose Cycle 2 Day 1: number analyzed (Participants) | 14
  Pre-dose Cycle 2 Day 1 | 326 (76.0)
  Pre-dose Cycle 2 Day 15: number analyzed (Participants) | 12
  Pre-dose Cycle 2 Day 15 | 216 (71.3)
  Pre-dose Cycle 3 Day 15: number analyzed (Participants) | 1
  Pre-dose Cycle 3 Day 15 | 87.7 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 4 Day 1: number analyzed (Participants) | 1
  Pre-dose Cycle 4 Day 1 | 87.6 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.

14. Secondary Outcome: Serum Trough Concentrations (Ctrough) of Amivantamab: on Day 1 of Cycle 3
Description: Ctrough of amivantamab at pre-dose on Day 1 of Cycle 3 were reported. Ctrough was defined as pre-dose serum drug concentration. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. As per change in planned analysis, data was not summarized for timepoint where number of participants analyzed were less than 3. Only individual participant data was available and reported.
Time Frame: Pre-dose at 0 hour on Day 1 of Cycle 3 (each cycle was of 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 2
mcg/mL
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 104 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 162 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.

15. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Amivantamab
Description: Terminal elimination half-life (t1/2) was the time measured for the serum concentration of a drug to decrease by half of its initial concentration. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: Pre-dose, 0, 2, 6, 24, 72, 168, 240 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 4
Hours | 201.3 (39.8)

16. Secondary Outcome: Accumulation Ratio (AR) of AUC (0-168 h) of Amivantamab
Description: Accumulation ratio for AUC was calculated as AUC (0-168 h) for Cycle 2 Day 1 divided by AUC (0-168 h) for Cycle 1 Day 1. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 4
Ratio | 2.85 (0.46)

17. Secondary Outcome: Number of Participants With Anti-Amivantamab Antibodies
Description: Number of participants with anti-amivantamab antibodies were reported. Serum samples were assessed for anti-drug antibodies.
Time Frame: From start of the treatment (Day 1) up to 30 days after the last dose of study drug (up to 3.8 months)
Population: Immunogenicity analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable postbaseline measurement. Here 'N' (overall number of participants analyzed) refers to the participants with appropriate samples had 1 or more samples obtained after their first amivantamab administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From screening up to 4.8 months; Serious AEs and Other AEs: From start of the treatment (Day 1) up to 30 days after last dose of study drug or start of subsequent anticancer therapy (up to 3.8 months)
Description: All treated analysis set included all participants who received at least 1 dose of study treatment.
Arm/Group | Amivantamab Monotherapy (1050/1400 mg)
All-Cause Mortality (participants affected / at risk) | 5/18
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amivantamab Monotherapy (1050/1400 mg) (N=18)
Ascites (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amivantamab Monotherapy (1050/1400 mg) (N=18)
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Eye Pain (Eye disorders) | 1
Eye Swelling (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Duodenal Ulcer (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 9
Alanine Aminotransferase Increased (Investigations) | 5
Aspartate Aminotransferase Increased (Investigations) | 5
Blood Alkaline Phosphatase Increased (Investigations) | 2
Blood Creatinine Increased (Investigations) | 1
Blood Glucose Increased (Investigations) | 2
Blood Urea Increased (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1
Glomerular Filtration Rate Decreased (Investigations) | 1
Prothrombin Time Prolonged (Investigations) | 1
Urinary Occult Blood (Investigations) | 1
Weight Decreased (Investigations) | 1
Weight Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 6
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 11
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT05653427/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05653427/SAP_001.pdf